CLINICAL TRIAL: NCT03296111
Title: Patients With Ocular Neuropathic Pain: Description of Pain and Impact on Their Quality of Life
Acronym: QUALVIDON
Status: Terminated | Type: Observational
Why Stopped: Difficulties for patients inclusion
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SDN_2017_9
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndromes; Neuralgia; Pain; Quality of Life
MeSH Terms: conditions — Dry Eye Syndromes; Neuralgia; Pain | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires on pain and quality of life — Patients will be asked to complete several questionnaires about their pain and the impact on their quality of life.
  They will complete the questionnaires in the ophthalmology consultation room or at home and return it by mail (or present it at the next consultation).
  Patients will be asked to complete several questionnaires :
  * Questionnaire about the characteristics of ocular neuropathic pain (7 items)
  * DEQ-5 (Dry Eye Questionnaire)
  * ODI (Ocular Surface Disease Index)
  * BPI (Brief Pain Inventory)
  * HADS (Hospital Anxiety and Depression Scale)

SUMMARY:
Some patients with dry eye may have severe disabling neuropathic pain. They describe spontaneous pain, dysesthesia, hyperalgesia or even allodynia. It is classical to note an important discordance between the high intensity of the symptoms and the poverty of the clinical signs. These pains are often unrecognized and therefore often not sufficiently treated. A significant impact on patient's quality of life may occur. The concept of ocular neuropathic pain being relatively recent, few studies have focused on the subject at present. Our study aims to shed light on these pains in patients consulting for dry eyes at the Ophthalmological Foundation A. de Rothschild.

The objective of our study is to describe precisely the characteristics of neuropathic eye pain and the visual, general and psychological repercussions in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older,
* Presenting at least one of the following symptoms: spontaneous pain, burning sensation in eye, dysesthesia, allodynia, hyperalgesia
* French language-skills

Exclusion Criteria:

* Severe corneal or palpebral damage explaining current pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ocular neuropathic pain.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Scores obtained with each questionnaires. | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtamologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No